CLINICAL TRIAL: NCT05440019
Title: Evaluation of the Safety and Usability of the M3T FERTIGO® System and Its Calibration
Brief Title: Evaluation of the Safety and Usability of the M3T Fertigo System and Its Calibration
Acronym: FERTIGO®
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-VLC-086-FC
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HEALTHY WOMEN IVI VALENCIA: Participants will be exposed to four sessions of image captures using FERTIGO® device.
  Prior to the session, a vaginal ultrasound (US) will be performed, for measuring the endometrial thickness as in the usual practice.
  Interventions: Device: IMAGE CAPTURE SESSION

INTERVENTIONS:
Device: IMAGE CAPTURE SESSION — The M3T FERTIGO® is an instrument to be used by a certified gynecologist and in particular by an IVF expert physician in order to observe and monitor the state of the endometrium lining of patients. The M3T device serves as a "mini hysteroscope" capable of magnification, capturing images and optional image processing thereof. The M3T enables to acquire in-vivo, magnified images of the endometrium surface, to identify key morphological parameters, calculate their attributes and statistics thereof and compare those for different acquisition images and to some "standard" tissue state tracks. One may then attempt to predict the Embryo transfer optimal timing, based on this analysis.

SUMMARY:
We have developed a new minimally invasive system for endometrial dating, that allows the physician to monitor, capture, project and analyze the actual morphology and maturity of the endometrial surface, at any given time. A time series of such indications provides an assessment regarding the pace of development by which the endometrium is maturing during a relevant cycle.

FERTIGO®'s method for endometrial dating has been validated in swine and ex-vivo human samples, where image analysis of tissues has been compared with traditional endometrial dating techniques. The comparison yielded calibration means and correlation between FERTIGO®'s dating and the traditional dating methods.

Thus, M3T FERTIGO®'s system is designed to enable the determination of the actual physiological cycle date, in good correlation with the indirect (endometrial thickness and hormones level) and delayed known methods (histopathology). To this end, a high quality, low magnification (X2-X4) image of the endometrium surface should be acquired, stored and analyzed.

This trial will evaluate, on the one hand, the safety and usability of the FERTIGO® device and, on the other hand, calibrate it by evaluating image quality. Both safety and usability will be measured through questionnaires answered by the participants (adverse events and satisfaction) and by the physicians (satisfaction), respectively, considering the introduction of the device, its use, and its removal.

ELIGIBILITY:
Inclusion criteria:

1. Healthy women
2. Age: 18 - 40, both inclusive
3. Regular menstrual cycles

Exclusion criteria:

1. Simultaneous participation in another clinical study that, at researcher's criteria, could interfere with the results of this study
2. Current pregnancy
3. Women with known existing endometrial pathology
4. Women with known oligo-ovulation or un-ovulation.
5. Women who were diagnosed with Endometriosis or Adenomyosis
6. Women with medical history of malignant tumors in their reproductive system
7. Women with IUD in place
8. Women menstruating on the day of the procedure
9. Women who have signs and symptoms of PID
10. Women who currently use any hormonal medications.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: The target population includes healthy women between 18 and 40 years with regular menstrual cycles.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and usability of the M3T for endometrium image capture | 1 month
  Measure of frequency and severity of all treatment-related adverse events, and physicians' satisfaction questionnaire

SECONDARY OUTCOMES:
To evaluate the captured image quality (calibration) | 1 month
  Measure the image quality.
To know the opinion/level of satisfaction of the study participants | 1 month
  Measure the satisfaction level of participants using questionaries

CONTACTS AND LOCATIONS:
Locations (1):
- Ivi Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
No decided jet